CLINICAL TRIAL: NCT04122001
Title: Transcranial Direct Current Stimulation in Typical and Atypical Alzheimer's Disease
Brief Title: Effects of Electrical Stimulation on Verbal Learning in Typical and Atypical Alzheimer's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00229164; 5R01AG068881 (NIH)
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease, Early Onset; Atypical Alzheimer's Disease; Logopenic Progressive Aphasia
Keywords: transcranial direct current stimulation (tDCS); Alzheimer's Disease (AD); verbal learning treatment; word list learning; logopenic Progressive Aphasia; episodic memory
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: This is a crossover design of active High-Definition tDCS (HD-tDCS) + Word List Learning Intervention (WordLLI) that crossovers to sham + WordLLI in Arm 1, and sham +WordLLI that crossovers to active HD-tDCS + WordLLI in Arm 2.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active HD-tDCS+word intervention then Sham+word intervention (Experimental): Participants will receive active HD-tDCS + Word List Learning Intervention (WordLLI) and then receive Sham + WordLLI after a three-month washout period.
  Interventions: Device: Active, in-person HD-tDCS or active remote tDCS; Device: Sham; Other: Word List Learning Intervention (WordLLI)
- Sham+word intervention then active HD-tDCS+word intervention (Experimental): Participants will receive Sham + Word List Learning Intervention (WordLLI) and then active HD-tDCS + WordLLI after a three-month washout period.
  Interventions: Device: Active, in-person HD-tDCS or active remote tDCS; Device: Sham; Other: Word List Learning Intervention (WordLLI)

INTERVENTIONS:
Device: Active, in-person HD-tDCS or active remote tDCS — Stimulation will be delivered by a battery-driven constant current stimulator. The electrical current will be administered to a pre-specified region of the brain (angular gyrus). The stimulation will be delivered at an intensity of 2 milliamperes (mA) (estimated current density 0.04 mA/cm2; estimated total charge 0.048 Coulombs/cm2) in a ramp-like fashion for a maximum of 20 minutes. In the active, in-person HD-tDCS the current is delivered in a ring configuration. In the active remote tDCS current is delivered in one electrode patch.
Device: Sham — Current will be administered in a ramp-like fashion but after the ramping the intensity will drop to 0 mA. Current under the Sham condition will last for a maximum of 30 seconds.
Other: Word List Learning Intervention (WordLLI) — Participants will receive a word list learning intervention (WordLLI) of semantically related and unrelated word lists. Word lists are presented across 10 trials, with an additional trial after a 10-minute delay to assess delayed recall. Immediately following verbal presentation of word lists during each trial, participants will be instructed to recall as many of the words from the list as possible. Participants may use the written modality as a strategy during recall. Word lists include 12 words matched based on psycholinguistics attributes (e.g., imageability, frequency). This task is designed to help participants improve memory via enhancing list learning capabilities.

SUMMARY:
Alzheimer's disease (AD) is the leading neurodegenerative disease of aging characterized by multiple cognitive impairments. Given the recent failures of disease-modifying drugs, the current focus is on preventing or mitigating synaptic damage that correlates with cognitive decline in AD patients. Transcranial Direct Current Stimulation (tDCS) is a safe, non-invasive, non-painful electrical stimulation of the brain that is shown to act as a primer at the synaptic level when administered along with behavioral therapy, mostly involving language, learning and memory. Previous studies have shown that tDCS over the left angular gyrus (AG) improves language associative learning in the elderly through changes in functional connectivity between the AG and the hippocampus. The investigators' previous clinical trial on the effects of tDCS in neurodegenerative disorders has also shown augmented effects of lexical retrieval for tDCS. In the present study the investigators will compare the effects of active vs. sham tDCS over the AG-an area that is part of the default mode network but also a language area, particularly important for semantic integration and event processing-in two predominant AD variants: probable AD with amnesic phenotype (amnesic/typical AD) and probable AD with non-amnesic (language deficit) phenotype also described as logopenic variant PPA with AD pathology (aphasic/atypical AD). The investigators aim to: (1) determine whether active high-definition tDCS (HD-tDCS) targeting the left AG combined with a Word-List Learning Intervention (WordLLI) will improve verbal learning; (2) identify the changes in functional connectivity between the stimulated area (AG) and other structurally and functionally connected areas using resting-state functional magnetic resonance imaging; (3) identify changes in the inhibitory neurotransmitter GABA at the stimulation site using magnetic resonance spectroscopy. Furthermore, the investigators need to determine the characteristics of the people that may benefit from the new neuromodulatory approaches. For this reason, the investigators will evaluate neural and cognitive functions as well as physiological characteristics such as sleep, and will analyze the moderating effects on verbal learning outcomes. Study results can help provide treatment alternatives as well as a better understanding of the therapeutic and neuromodulatory effects of tDCS in AD, thus improving patients' and caregivers' quality of life.

DETAILED DESCRIPTION:
The investigation implements a double-blind, sham-controlled, within-subject, cross-over design that allows for the evaluation of the cognitive and neural effects of word-list learning as modulated by tDCS compared to sham stimulation. Participants in all groups will receive word-list learning intervention (WordLLI)+ High-Definition tDCS (HD-tDCS) or WordLLI+ sham in Period 1 or 2, randomized for the Period 1 stimulation condition. Each learning Period will last 2 weeks, with 5 learning sessions per week (for a total of 10 learning sessions per Period) with a 3-month (stimulation-free) wash-out period between the two Periods. The intensity, total number of learning sessions and number of learning items is consistent with most other tDCS studies in neurodegenerative disorders and the investigators have used this design successfully over the past 7 years in neurodegenerative disorders (PPA, mild AD). Stimulation is implemented every weekday to take advantage of the long-term potentiation induced by tDCS as found in early multi-session studies. A tDCS-only condition (without any intervention) is not implemented in this design because no study to date has shown improvement on motor, cognitive, or language performance after anodal tDCS-only for 2 or even more weeks. After each period the investigators will perform 1-month and 3-month follow-up sessions for evaluation purposes. For those participants who are long-distance, at the 1-month time point only the investigators may use a video conferencing tool such as GoToMeeting to administer the assessments. This is to mitigate the costs of travel for a short appointment.

ELIGIBILITY:
Inclusion Criteria:

For the aphasic/atypical AD participants:

* Must be between 45-85 years of age.
* Must be right-handed.
* Must be proficient in English.
* Must have a minimum of high-school education.
* Must be diagnosed as logopenic variant Primary Progressive Aphasia (PPA) with Alzheimer's Disease (AD) biomarkers. Other possible diagnosis for the 'aphasic AD' variant would be Mild Cognitive Impairment (MCI) or 'possible AD' according to 2011 guidelines with AD biomarkers (CSF or positron emission tomography (PET) amyloid-beta or fluorodeoxyglucose (FDG)-positron emission tomography (PET) with unihemispheric atrophy).
* Participants will be diagnosed from PPA and early dementias clinics at Johns Hopkins University or other specialized centers in US using current consensus criteria. Diagnosis will be based on neuropsychological testing, language testing (most commonly the Western Aphasia Battery), MRI and clinical assessment. The investigators will also use two new variant classification tests the investigators have developed at the lab which discriminate PPA variants with great accuracy (above 80%): a spelling test and a speech production test (i.e.,Cookie Theft picture description task).

For the amnesic/typical AD participants:

* Must be between 45-85 years of age.
* Must be right-handed.
* Must be proficient in English.
* Must have a minimum of high-school education.
* Must be diagnosed with 'probable AD' in specialized diagnostic centers with neuropsychological (e.g., RAVLT) and AD biomarkers according to 2011 guidelines.
* The investigators will also perform extensive testing in the investigators' test battery including the Mnemonic Similarity Test (MST) that discriminates and measures the most salient hippocampal deficit-pattern separation (PS).

Exclusion Criteria:

* People with previous neurological disease including vascular dementia (e.g., stroke, developmental dyslexia, dysgraphia or attentional deficit).
* People with hearing loss (> 25 decibel, using audiometric hearing screen).
* People with uncorrected visual acuity loss.
* People with advanced dementia or severe language impairments (MMSE < 15, or Montreal Cognitive Assessment <10, or language Frontotemporal Dementia-specific Clinical Dementia Rating (FTD-CDR) = 3).
* Left handed individuals.
* People with pre-existing psychiatric disorders such as behavioral disturbances, severe depression, or schizophrenia that do not allow these people to comply or follow the study schedule and requirements such as repeated evaluation and therapy.

Exclusion Criteria for MRI Participation:

* People with severe claustrophobia.
* People with cardiac pacemakers or ferromagnetic implants.
* Pregnant women.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-08-17 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in auditory recall accuracy based on the sum of words recalled in Trials 1-5 of semantically related - trained word-lists | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Each trained word-list (practiced during the intervention period) will consist of 12 semantically related words (e.g., birds). Word lists will be constructed using psycholinguistic databases. There will be 5 Trials to learn each list. The investigators will compute the raw score of items correctly recalled by summing all scores from Trial 1 to Trial 5 and transforming to percent correct (range: 0-100%) at each time point of the study. Increase in scores is considered a benefit.
Change in auditory delayed recall accuracy of semantically related - trained word-lists | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Each trained word-list (practiced during the intervention period) will consist of 12 semantically related words (e.g., birds). Word lists will be constructed using psycholinguistic databases. There will be 5 Trials to recall each list, and then participants will be asked to recall that list 20 minutes later (delayed recall). The investigators will compute the raw score of items correctly recalled (delayed recall) and transform to percent correct (range: 0-100%) at each time point of the study. Increase in scores is considered a benefit.
Change in auditory recall accuracy based on the sum of words recalled in Trials 1-5 of semantically unrelated - trained word-lists | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Each trained word-list (practiced during the intervention period) will consist of 12 semantically unrelated words (as in RAVLT). Word lists will be constructed using psycholinguistic databases. There will be 5 Trials to learn each list. The investigators will compute the raw score of items correctly recalled by summing all scores from Trial 1 to Trial 5 and transforming to percent correct (range: 0-100%) at each time point of the study. Increase in scores is considered a benefit.
Change in auditory delayed recall accuracy of semantically unrelated - trained word-lists | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Each trained word-list (practiced during the intervention period) will consist of 12 semantically unrelated words (as in RAVLT). Word lists will be constructed using psycholinguistic databases. There will be 5 Trials to recall each list, and then participants will be asked to recall that list 20 minutes later (delayed recall). The investigators will compute the raw score of items correctly recalled (delayed recall) and transform to percent correct (range: 0-100%) at each time point of the study. Increase in scores is considered a benefit.
Change in auditory recall accuracy based the sum of words recalled in Trials 1-5 of semantically related - untrained word-lists | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Each untrained word-list (not practiced during the intervention period) will consist of 12 semantically related words (e.g., birds). Word lists will be constructed using psycholinguistic databases. There will be 5 Trials to learn each list. The investigators will compute the raw score of items correctly recalled by summing all scores from Trial 1 to Trial 5 and transforming to percent correct (range: 0-100%) at each time point of the study. Increase in scores is considered a benefit.
Change in auditory delayed recall accuracy of semantically related - untrained word-lists | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Each untrained word-list (not practiced during the intervention period) will consist of 12 semantically related words (e.g., birds). Word lists will be constructed using psycholinguistic databases. There will be 5 Trials to recall each list, and then participants will be asked to recall that list 20 minutes later (delayed recall). The investigators will compute the raw score of items correctly recalled (delayed recall) and transform to percent correct (range: 0-100%) at each time point of the study. Increase in scores is considered a benefit.
Change in auditory recall accuracy based on the sum of words recalled in Trials 1-5 of semantically unrelated - untrained word-lists | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Each untrained word-list (not practiced during the intervention period) will consist of 12 semantically unrelated words (as in RVLT). Word lists will be constructed using psycholinguistic databases. There will be 5 Trials to learn each list. The investigators will compute the raw score of items correctly recalled by summing all scores from Trial 1 to Trial 5 and transforming to percent correct (range: 0-100%) at each time point of the study. Increase in scores is considered a benefit.
Change in auditory delayed recall accuracy of semantically unrelated - untrained word-lists | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Each untrained word-list (not practiced during the intervention period) will consist of 12 semantically unrelated words (as in RVLT). Word lists will be constructed using psycholinguistic databases. There will be 5 Trials to recall each list, and then participants will be asked to recall that list 20 minutes later (delayed recall). The investigators will compute the raw score of items correctly recalled (delayed recall) and transform to percent correct (range: 0-100%) at each time point of the study. Increase in scores is considered a benefit.

SECONDARY OUTCOMES:
Change in Rey Auditory-Verbal Learning Test (RAVLT) score | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  RAVLT is a well-established verbal memory test. RAVLT includes a 5-trial presentation of a 15-word list (List A), a single presentation of an interference list (List B)(Trial 6), two post-interference recall trials (one immediate - Trial 7, one delayed - Trial 8) and recognition of the target words in the orthographic modality with distractors (Trial 9). Scoring includes the percent score of Trial 1, Trial 5, Trial 8 and Trial 9 as well as the sum of Trial 1 through 5, and the difference between Trial 5 and Trial 1 computed as the percent difference between the scores before intervention and each time point after. Increase in score is considered a benefit.
Change in Mini Mental State Examination (MMSE) | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  MMSE is a well-established cognitive assessment test. It examines functions including registration (repeating named prompts), attention and calculation, recall, language, ability to follow simple commands and orientation. The total raw score is out of 30 points. The investigators will compute the raw score of items correct and transform to percent correct (range: 0-100%), computing change in outcome in percent difference between before intervention and each time point after. Increase in score is considered a benefit.
Change in Mnemonic Similarity Task (MST) score | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  MST is a well-established test in order to assess high interference memory and general recognition memory via pattern separation. It involves differentiating between previously learned images and novel images. For the MST tasks, the Pattern Separation (PS) score will be calculated using two measures: a) the rate of similar items correctly identified minus the rate of similar items misidentified as new (S|S-S|N); b) the rate of similar items correctly identified minus the rate of similar items misidentified as old (S|S-O|S). The number of correct responses for each category of items (i.e., old, similar, new) and the type of errors (i.e., identifications of new items as similar; identification of similar items as old) will also be tracked. Change in outcome in percent difference will be computed between the scores before intervention and each time point after. Increase in scores is considered a benefit.
Change in word repetition score | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Temple Assessment of Language and Short-Term Memory in Aphasia (TALSA) tasks include word repetition, with sets of 1-6 words. Scoring will be based on percent of words correctly repeated. The investigators will compute the raw score of items correct and transform to percent correct (range: 0-100%), computing change in outcome in percent difference between before intervention and each time point after. Increase in score is considered a benefit.
Change in non-word repetition score | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  TALSA tasks include non-word repetition, with sets of 1-6 non-words. Scoring will be based on percent of non-words correctly repeated. The investigators will compute the raw score of items correct and transform to percent correct (range: 0-100%), computing change in outcome in percent difference between before intervention and each time point after. Increase in score is considered a benefit.
Change in sentence repetition score | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Sentence repetition tasks come from the TALSA, with scoring based on percent of words in sentences correctly repeated. The investigators will compute the raw score of items correct and transform to percent correct (range: 0-100%), computing change in outcome in percent difference between before intervention and each time point after. Increase in score is considered a benefit.
Change in oral naming Boston Naming Test score | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Accuracy in oral picture naming (30-item Boston Naming Test) will be compared for tDCS and sham conditions. The Boston Naming Test is a widely used picture naming test that detects lexical retrieval deficits in the oral modality. The investigators will compute the raw score of items correct and transform to percent correct (range: 0-100%), computing change in outcome in percent difference between before intervention and each time point after. Increase in score is considered a benefit.
Change in oral naming Philadelphia Naming Test score | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Accuracy in oral picture naming (Philadelphia Naming Test) will be compared for tDCS and sham conditions. The Philadelphia Naming Test is an extensive picture naming test that comprises 275 items from a wide range of frequencies and other psycholinguistic characteristics. The investigators will compute the raw score of items correct and transform to percent correct (range: 0-100%), computing change in outcome in percent difference between before intervention and each time point after. Increase in score is considered a benefit.
Change in written naming as assessed by Boston Naming Test | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Accuracy in written picture naming (30-item Boston Naming Test) will be compared for tDCS and sham conditions. The investigators will compute the raw score of items correct and transform to percent correct (range: 0-100%), computing change in outcome in percent difference between before intervention and each time point after. Increase in score is considered a benefit.
Change in written naming as assessed by Philadelphia Naming Test | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Accuracy in written picture naming (Philadelphia Naming Test) will be compared for tDCS and sham conditions. The investigators will compute the raw score of items correct and transform to percent correct (range: 0-100%), computing change in outcome in percent difference between before intervention and each time point after. Increase in score is considered a benefit.
Change in oral naming of action as assessed by Hopkins Assessment of Naming Actions (HANA) | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Accuracy in oral naming of actions will be compared for tDCS and sham conditions. The investigators will compute the raw score of items correct and transform to percent correct (range: 0-100%), computing change in outcome in percent difference between before intervention and each time point after. Increase in score is considered a benefit.
Change in syntactic comprehension as assessed by Subject-relative, Object-relative, Active, Passive (S.O.A.P.) Syntactic Battery | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  The 40-item Subject-relative, Object-relative, Active, Passive (S.O.A.P.) Syntactic Battery of various sub-tests will be used to assess argument structure comprehension and production. The investigators will compute the raw score of items correct and transform to percent correct (range: 0-100%), computing change in outcome in percent difference between baseline and each time point. Increase in score is considered benefit.
Change in verbal fluency task score | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Verbal fluency tasks (semantic and letter fluency) involve generating as many words as possible in one minute. Scoring will be based on number of words generated per minute. The investigators will compute the raw score of items correct and compute change in outcome between baseline and each time point. Increase in score is considered benefit.
Change in spelling as assessed by the Johns Hopkins Dysgraphia battery | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Accuracy in spelling using the Johns Hopkins Dysgraphia battery will be compared for tDCS and sham conditions. The investigators will compute the raw score of items correct using a spelling scoring system accounting for additions, substitutions, and deletions, and transform to percent correct (range: 0-100%), computing change in outcome in percent difference before intervention and each time point after. Increase in score is considered a benefit.
Change in digit span forward score | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Digit span forward involves the recall of a series of single digits (sets of 1-8 digits) in the same order the digits were presented. Scoring will be based on the number of consecutive digits correctly recalled. The investigators will compute the change in outcome between the time point before intervention and each time point after. Increase in score is considered a benefit.
Change in digit span backward score | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Digit span backward involves the recall of a series of single digits (sets of 1-8 digits) in the reverse order than the digits were presented. Scoring will be based on the number of consecutive digits correctly recalled. The investigators will compute the change in outcome between the time point before intervention and each time point after. Increase in score is considered a benefit.
Change in spatial span forward score | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Spatial span forward involves the recall of a series of positions on a board (sets of 1-9) in the same order the digits were presented. Scoring will be based on the number of consecutive positions correctly recalled. The investigators will compute the change in outcome between the time point before intervention and each time point after. Increase in score is considered a benefit.
Change in spatial span backward score | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Spatial span backward involves the recall of a series of positions (sets of 1-8) in the reverse order than the digits were presented. Scoring will be based on the number of consecutive positions correctly recalled. The investigators will compute the change in outcome between the time point before intervention and each time point after. Increase in score is considered a benefit.
Change in semantic content of connected speech | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Using the Cookie Theft image from the Boston Diagnostic Aphasia Examination (BDAE) and the Circus image from the Apraxia Battery for Adults (ABA) investigators will obtain representative language samples as participants describe the images. The investigators will compute the raw score of items (semantics) correct and transform to percent correct (range: 0-100%), computing change in outcome in percent difference between before intervention and each time point after. Increase in score is considered a benefit.
Change in attention and manipulation of information scores | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Using the Trail Making Test (TMT) parts A and B, which include the sequential connection of letters/numbers in order to complete a trail, the investigators will obtain the time required by the participants to finish the tasks. Decrease in the time is considered a benefit.
Change in volumetric measurements of select brain regions | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Using Magnetization-Prepared Rapid Gradient-Echo (MPRAGE) Magnetic Resonance Imaging (MRI) investigators will perform volumetric measurements of select brain regions. Measurements will be collected in millimeters cubed (mm^3).
Change in functional connectivity of select brain regions (z-correlations) | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Using resting stage functional MRI (rs-fMRI) investigators will detect activity of various brain regions under a resting/task-negative condition, which will help evaluate functional regional interactions as indicated by the z-correlations between the selected brain area.
Change in Gamma-Aminobutyric Acid (GABA) concentration | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Using Magnetic Resonance Spectroscopy (MRS) investigators will measure metabolite (GABA) concentrations from select brain regions in international units (IU).
Change in location of white matter tracts of select brain regions | Before intervention, immediately after intervention, 1 month and 3 months post intervention, up to 31 weeks
  Using Diffusion Tensor Imaging (DTI) investigators will estimate the location of the brain's white matter tracts on the regions of concern.
Change in anisotropy of white matter tracts of select brain regions | Before intervention, immediately after intervention and 3 months post intervention, up to 31 weeks
  Using Diffusion Tensor Imaging (DTI) investigators will estimate the anisotropy of the brain's white matter tracts on the brain regions of concern.

OTHER OUTCOMES:
Correlation of primary and secondary outcomes with sleep efficiency | One week before intervention and one week post intervention, up to 8 weeks
  Actigraphy for sleep is a method for observing sleep activity patterns. Actigraphy data is gathered via a wrist band with an accelerometer and a light detector. The investigators will compute the sleep efficiency (% of time in bed spent asleep) and assess whether it correlates with the performance on primary or secondary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Kyrana Tsapkini, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsapkini K, Frangakis C, Gomez Y, Davis C, Hillis AE. Augmentation of spelling therapy with transcranial direct current stimulation in primary progressive aphasia: Preliminary results and challenges. Aphasiology. 2014;28(8-9):1112-1130. doi: 10.1080/02687038.2014.930410. PMID 26097278
- [Background] Tsapkini K, Webster KT, Ficek BN, Desmond JE, Onyike CU, Rapp B, Frangakis CE, Hillis AE. Electrical brain stimulation in different variants of primary progressive aphasia: A randomized clinical trial. Alzheimers Dement (N Y). 2018 Sep 5;4:461-472. doi: 10.1016/j.trci.2018.08.002. eCollection 2018. PMID 30258975
- [Background] Ficek BN, Wang Z, Zhao Y, Webster KT, Desmond JE, Hillis AE, Frangakis C, Vasconcellos Faria A, Caffo B, Tsapkini K. The effect of tDCS on functional connectivity in primary progressive aphasia. Neuroimage Clin. 2018 May 21;19:703-715. doi: 10.1016/j.nicl.2018.05.023. eCollection 2018. PMID 30009127
- [Background] Reis J, Schambra HM, Cohen LG, Buch ER, Fritsch B, Zarahn E, Celnik PA, Krakauer JW. Noninvasive cortical stimulation enhances motor skill acquisition over multiple days through an effect on consolidation. Proc Natl Acad Sci U S A. 2009 Feb 3;106(5):1590-5. doi: 10.1073/pnas.0805413106. Epub 2009 Jan 21. PMID 19164589
- [Background] Huey ED, Probasco JC, Moll J, Stocking J, Ko MH, Grafman J, Wassermann EM. No effect of DC brain polarization on verbal fluency in patients with advanced frontotemporal dementia. Clin Neurophysiol. 2007 Jun;118(6):1417-8. doi: 10.1016/j.clinph.2007.02.026. Epub 2007 Apr 23. No abstract available. PMID 17452012
- [Background] Antal A, Terney D, Poreisz C, Paulus W. Towards unravelling task-related modulations of neuroplastic changes induced in the human motor cortex. Eur J Neurosci. 2007 Nov;26(9):2687-91. doi: 10.1111/j.1460-9568.2007.05896.x. Epub 2007 Oct 26. PMID 17970738
- [Background] Segrave RA, Arnold S, Hoy K, Fitzgerald PB. Concurrent cognitive control training augments the antidepressant efficacy of tDCS: a pilot study. Brain Stimul. 2014 Mar-Apr;7(2):325-31. doi: 10.1016/j.brs.2013.12.008. Epub 2013 Dec 19. PMID 24486425
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Background] Gorno-Tempini ML, Hillis AE, Weintraub S, Kertesz A, Mendez M, Cappa SF, Ogar JM, Rohrer JD, Black S, Boeve BF, Manes F, Dronkers NF, Vandenberghe R, Rascovsky K, Patterson K, Miller BL, Knopman DS, Hodges JR, Mesulam MM, Grossman M. Classification of primary progressive aphasia and its variants. Neurology. 2011 Mar 15;76(11):1006-14. doi: 10.1212/WNL.0b013e31821103e6. Epub 2011 Feb 16. PMID 21325651
- [Background] Neophytou K, Wiley RW, Rapp B, Tsapkini K. The use of spelling for variant classification in primary progressive aphasia: Theoretical and practical implications. Neuropsychologia. 2019 Oct;133:107157. doi: 10.1016/j.neuropsychologia.2019.107157. Epub 2019 Aug 8. PMID 31401078
- [Background] Riello M, Faria AV, Ficek B, Webster K, Onyike CU, Desmond J, Frangakis C, Tsapkini K. The Role of Language Severity and Education in Explaining Performance on Object and Action Naming in Primary Progressive Aphasia. Front Aging Neurosci. 2018 Oct 30;10:346. doi: 10.3389/fnagi.2018.00346. eCollection 2018. PMID 30425638